CLINICAL TRIAL: NCT04915651
Title: Prospective Study of Gallbladder Cryoablation in High-Risk Surgical Patients
Brief Title: Gallbladder Cryoablation in High-Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Hugh McGregor, Associate Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1904567382
Record Dates: First submitted 2021-05-28; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Gallbladder Diseases; Cholecystitis; Biliary Colic; Gallstone; Cholecystitis; Biliary Dyskinesia; Gallstone; Gall Bladder Pain
Keywords: cryoablation; gallstones; gallbladder; cholecystitis
MeSH Terms: conditions — Gallbladder Diseases; Cholecystitis; Acalculous Cholecystitis; Biliary Dyskinesia; Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Gallbladder Cryoablation (Experimental): High-risk patients who undergo gallbladder cryoablation
  Interventions: Device: Gallbladder Cryoablation

INTERVENTIONS:
Device: Gallbladder Cryoablation — Percutaneous cryoablation of the gallbladder.

SUMMARY:
Benign gallbladder disease, including acute cholecystitis, chronic cholecystitis, biliary dyskinesia, and biliary colic, is very common, with over 300,000 surgical cholecystectomies performed per year in the US. Unfortunately, complication rates in elderly patients or patients with many comorbidities are high. These patients are often managed with percutaneous tube drainage of the gallbladder (percutaneous cholecystostomy). The recurrence rate of calculous cholecystitis after cholecystostomy tube removal is as high as 35% at 1 year. These patients are thus faced with permanent cholecystostomy tube drainage, high-risk surgery, or cholecystostomy tube removal and risk of repeat cholecystitis. Gallbladder cryoablation is an alternative to surgical cholecystectomy which is performed percutaneously and does not require general anesthesia. Published evidence on the outcomes of gallbladder cryoablation is however limited at this point in time. The purpose of the proposed study is to follow the outcomes of high-risk patients who undergo gallbladder cryoablation.

DETAILED DESCRIPTION:
The purpose of the proposed research is to evaluate the outcomes of gallbladder cryoablation in high-risk surgical candidates with benign gallbladder disease (acute cholecystitis, chronic cholecystitis, biliary dyskinesia, biliary colic).

Specific Aim:

Aim 1: To evaluate the safety and efficacy of gallbladder cryoablation in high-risk surgical candidates. Patients who undergo gallbladder cryoablation will be followed long-term according to standard of care. This includes scheduled clinic follow up, laboratory analysis, and imaging as needed. We hypothesize that gallbladder cryoablation is a safe and effective treatment for high-risk surgical patients with benign gallbladder disease. Clinically, we hypothesize that patients will be free from any clinical symptoms or signs after gallbladder cryoablation and removal of a cholecystostomy tube. These include, but are not limited to right upper quadrant pain, fever, chills, and jaundice.

Aim 2: To evaluate the imaging changes seen in the gallbladder after cryoablation. Imaging is part of routine follow up after percutaneous ablation and may include CT, MRI, and nuclear medicine studies as needed. We hypothesize that after cryoablation, patients will be functionally acholecystic, which occlusion of the cystic duct and involution and fibrosis of the gallbladder demonstrated by imaging.

ELIGIBILITY:
Inclusion Criteria:

* High-risk surgical candidates with benign gallbladder disease who are not eligible for surgical cholecystectomy and are able to consent to study inclusion.

Exclusion Criteria:

* Patients with benign gallbladder disease who are eligible for surgical cholecystectomy or who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Symptomatic relief | Up to 2 years after procedure
  Absence of right upper quadrant abdominal pain and nausea and absence of repeat episodes of cholecystitis, which would manifest as right upper quadrant abdominal pain associated with a fever (>100 C) and leukocytosis.
Complications | Up to 2 years after procedure
  Clavien-Dindo classification complications

SECONDARY OUTCOMES:
Imaging | Up to 2 years after procedure
  Imaging evidence of gallbladder devitalization and fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Hugh McGregor, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No